CLINICAL TRIAL: NCT01818908
Title: A Prospective, Single-arm, Open-label, Phase 2 Study to Evaluate Efficacy and Safety of DA-EPOCH Regimen for Non-Hodgkin's Lymphoma With Hemophagocytic Lymphohistiocytosis
Brief Title: Trial of DA-EPOCH Regimen for NHL With HLH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-HLH-001
Record Dates: First submitted 2013-03-23; First posted 2013-03-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: NHL With Hemophagocytic Lymphohistiocytosis
Keywords: non-Hodgkin's lymphoma; hemophagocytic lymphohistiocytosis; DA-EPOCH; rituximab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphohistiocytosis, Hemophagocytic | interventions — EPOCH protocol; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DA-EPOCH (Experimental): Infused agents:
  Etoposide 50 mg/m2/day CI24h d1-d4; Doxorubicin 10 mg/m2/day CI24h d1-d4; Vincristine 0.4mg/m2/day CI24h d1-d4;
  Bolus agents:
  Rituximab(B-NHL) 375 mg/m2/day IV d0; Cyclophosphamide 750 mg/m2/day IV d5 ; Prednisone 60 mg/m2/bid oral or IV d1-d5;
  The details of dose adjustment are described in ref 1.
  If enrolled patient was histologically confirmed CD20+ B cell lymphoma, standard dose of rituximab will be recommend to combined with DA-EPOCH regimen.
  Interventions: Drug: DA-EPOCH

INTERVENTIONS:
Drug: DA-EPOCH — DA-EPOCH regimen
  Other Names: Infused agents; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone; Rituximab(B-NHL)

SUMMARY:
The major purpose of this clinical study is to assess clinical outcome of dose-adjusted EPOCH regimen for patients with non-Hodgkin's lymphoma(NHL)-associated hemophagocytic lymphohistiocytosis

DETAILED DESCRIPTION:
Lymphoma-associated hemophagocytic lymphohistiocytosis(LA-HLH) has a high fatality rate and the worst outcome. The major cause of LA-HLH is aggressive non-Hodgkin's lymphoma(NHL), especially T/NKT cell lymphomas. Until now, there is no recommended therapeutic schedule for this fatal disease. Dose-adjusted(DA) EPOCH (etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin) shows effective activity in patients with aggressive NHL, which also contains the critical drugs for HLH of HLH-94/04. The investigators therefore developed DA-EPOCH regimen to treat non-Hodgkin's lymphoma with hemophagocytic lymphohistiocytosis and assess its clinical outcome including safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1 .Histologically confirmed non-Hodgkin's lymphoma; 2. Patients whose clinical findings satisfy either of HLH 2004 standard: 3. newly-diagnosed and untreated; 4. understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements.

HLH2004 standard at least 5 criteria out of the following: Fever ≥ 38.5 ℃ for ≥ 7 days; hepatosplenomegaly; Cytopenias affecting ≥ 2 of 3 lineages in PB Hb < 9 g/L Platelet < 100 x 109 /L ANC < 1.0 x 109 /L; Hypertriglyceridemia and/or hypofibrinogenemia (fasting triglycerides ≥ 265 mg/dL, fibrinogen ≤ 1.5 g/L); Hemophagocytosis in BM or spleen or LN; Low or absent NK-cell activity ( according to local laboratory reference); Serum-ferritin ≥ 500 mcg/L ; Soluble CD25(sIL-2 receptor) ≥ 2,400 U/ml ; 3.New-diagnosed and untreated; 4.Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements.

Exclusion criteria

1. primary HLH;
2. HLH from rheumatic disorder (such as systemic Lupus Erythematosus, adult onset still disease, antiphospholipid antibody syndrome);
3. pregnancy (as determined by serum or urine test) or active breast feeding;
4. concomitant malignancy other than NHL and need to treat;
5. concomitant with other hematologic diseases (such as leukemia, hemophilia primary myelofibrosis) which investigators considered it unsuitable to be enrolled into this clinical trial;
6. any potential drug abuse, medical, psychological or social conditions which may disturb this investigation and assessment;
7. in any conditions which investigator considered ineligible for this study

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2018-10 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
overall response rate | one year
  overall response rate after treated by DA-EPOCH regimen

SECONDARY OUTCOMES:
progression free survival | one year
  progression free survival after treatment of DA-EPOCH regimen
overall survival | one year
  overall survival after treatment of DA-EPOCH regimen
Number of Participants with Adverse Events | up to 30 days after last dose of treatment
  Number of Participants with Adverse Events, and evaluated standard is according to common terminology criteria adverse events(CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (4):
- China (4):
  - ChangZhou No.2 People's Hospital, Changzhou, Jiangsu
  - HuaiAn First People's Hospital, HuaiAn, Jiangsu
  - JiangSu Province Hospital, Nanjing, Jiangsu
  - WuXi People's Hospital, Wuxi, Jiangsu

REFERENCES:
- [Background] Wilson WH, Grossbard ML, Pittaluga S, Cole D, Pearson D, Drbohlav N, Steinberg SM, Little RF, Janik J, Gutierrez M, Raffeld M, Staudt L, Cheson BD, Longo DL, Harris N, Jaffe ES, Chabner BA, Wittes R, Balis F. Dose-adjusted EPOCH chemotherapy for untreated large B-cell lymphomas: a pharmacodynamic approach with high efficacy. Blood. 2002 Apr 15;99(8):2685-93. doi: 10.1182/blood.v99.8.2685. PMID 11929754
- [Background] Henter JI, Horne A, Arico M, Egeler RM, Filipovich AH, Imashuku S, Ladisch S, McClain K, Webb D, Winiarski J, Janka G. HLH-2004: Diagnostic and therapeutic guidelines for hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2007 Feb;48(2):124-31. doi: 10.1002/pbc.21039. PMID 16937360
- [Background] Wilson WH, Dunleavy K, Pittaluga S, Hegde U, Grant N, Steinberg SM, Raffeld M, Gutierrez M, Chabner BA, Staudt L, Jaffe ES, Janik JE. Phase II study of dose-adjusted EPOCH and rituximab in untreated diffuse large B-cell lymphoma with analysis of germinal center and post-germinal center biomarkers. J Clin Oncol. 2008 Jun 1;26(16):2717-24. doi: 10.1200/JCO.2007.13.1391. Epub 2008 Mar 31. PMID 18378569